CLINICAL TRIAL: NCT07269613
Title: Comparison of Ultrasound Guided Pulsed Radiofrequency Versus Hyaluronidase Hydrodissection for Treatment of Carpal Tunnel Syndrome, a Prospective, Randomized, Controlled Clinical Study
Brief Title: Pulsed Radiofrequency Versus Hyaluronidase Hydrodissection for Treatment of Carpal Tunnel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amany Mahmoud Mohamed, Resident of Anesthesia, ICU and Pain management faculty of medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-25-9-20MS
Record Dates: First submitted 2025-09-29; First posted 2025-12-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: pulsed radiofrequency versus hyaluronidase hydrodissection for treatment of carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (PRF Group) (Active Comparator): Group A (PRF Group): will Receive ultrasound-guided pulsed radiofrequency to the median nerve at the carpal tunnel.
  Interventions: Procedure: Pulsed Radiofrequency
- Group B (HD Group) (Active Comparator): Group B (HD Group): will Receive ultrasound-guided hydrodissection of the median nerve using hyaluronidase solution.
  Interventions: Procedure: Hyaluronidase Hydrodissection

INTERVENTIONS:
Procedure: Pulsed Radiofrequency — Pulsed Radiofrequency:
  Top neuropole needle 100-mm with a 10-mm active tip will be advanced with
  ultrasound guidance using the in-plane technique towards the median nerve.
  Sensory and motor stimulation will be tested when the needle is close to the median nerve.
  During sensory stimulation (50 Hz; 1-ms pulsed width; 0-3.0 volt), the patients will report paresthesia in the distal fingers.
  After performing a motor stimulation (2 Hz; 1-ms pulsed width; 0-3.0 volt), contractions of the thenar muscle will be observed.
  PRF lesion will then be carried out for 6 min, pulse width of 5 MS, 5 pulses per second and 35 volts at 42°C.
  Arms: Group A (PRF Group)
Procedure: Hyaluronidase Hydrodissection — Hyaluronidase Hydrodissection:
  The patient will sit facing the examiner with the forearm supinated and semiflexed at 90°, and the wrist placed on the examination couch with semi extended fingers. The injection for a 5 mL volume of HD 1500 IU will be done under complete sterile conditions. A 26-gauge needle will be introduced from the lateral side toward the midline, using the in-plane approach to target the median nerve in the carpal tunnel using the ulnar approach.
  Ultrasonographic visualization of the needle tip will be continuous, the injection was done gradually, and the needle will be advanced dissecting the flexor retinaculum away from the median nerve via gradual drug infiltration.
  Arms: Group B (HD Group)

SUMMARY:
The aim of this study is to compare the clinical efficacy and safety of ultrasound-guided pulsed radiofrequency and hyaluronidase hydrodissection in the treatment of carpal tunnel syndrome. This research seeks to evaluate both techniques in terms of pain relief, functional improvement, nerve conduction parameters, and potential complications, in order to identify the more effective minimally invasive approach for managing carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20-80 years
2. Clinical diagnosis of CTS with symptoms for at least 3 months
3. Electrophysiological evidence of mild to moderate CTS
4. No previous intervention for CTS in the affected hand

Exclusion Criteria:

1. Previous wrist surgery or trauma
2. Medical history of polyneuropathy, thoracic outlet syndrome, or brachial plexopathy
3. Coagulopathy or local infection at injection site
4. Pregnancy or breastfeeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Onset time of significant pain relief | 1 month
  The VAS will be used to quantify pain on the scale of 0 (no pain) to 10 (extremely severe pain). Onset time will be defined as the day when the VAS score declined by 40% or more

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | 1 week and 1, 3, 6 months
  BCTQ is the most used questionnaire in clinical studies for evaluation of the symptom severity and functional status of patients with CTS [9]. Symptom severity is rated based on 11 questions scored from 1 point (mildest) to 5 points (most severe), and the functional status is evaluated with 8 questions scored from 1 point (no difficulty with activity) to 5 points (cannot perform the activity at all)
Cross-sectional area (CSA) | baseline and then at 1-, 3-, and 6-months
  CSA of the median nerve will be measured at the proximal inlet of the carpal tunnel (at the level of the pisiform bone) by the same physician. The patients hold their wrists in a neutral position with the palm up and the fingers semi-extended. CSA will be measured three times, and the mean will be used for the analysis. Typically, a CSA greater than 9-10 mm2 at the wrist is considered suggestive of carpal tunnel syndrome. The ultrasonographic evaluation of median nerve CSA has high sensitivity (89%) and specificity (83%) for the diagnosis of CTS.
  This will be done at baseline and then at 1-, 3-, and 6-months post-injection. All measurements will be performed three times, and the mean of the three measurements was used for further statistical analyses
Sensory nerve conduction velocity (SNCV) | baseline and 1, 3, and 6months post-injection
  The antidromic SNCV of the median nerve will be measured in all subjects. All examinations will be performed by the same physician in the same room maintained at a constant temperature of 25°C. Skin temperature on the hand and wrist will be maintained between 32.0 and 34.0°C. Active and reference ring electrodes will be placed over the 2nd proximal and distal interphalangeal joints. The median nerve will be stimulated at the wrist between the palmar longus and flexor carpal radialis tendon at approximately 14 cm from the active electrode. will performed at baseline and 1, 3, and 6months post-injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided